CLINICAL TRIAL: NCT05726123
Title: Physiological and Functional Effects of Therapeutic Intervention With Neuromodulation Suit With and Without Combination of Reverse Virtual Reality in Fibromyalgia Patients.
Brief Title: Therapeutic Intervention With Neuromodulation and Inverse Virtual Reality in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Clinical Proffesor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 28922
Record Dates: First submitted 2023-01-19; First posted 2023-02-13 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Fibromyalgia
Keywords: neuromodulation; fibromyalgia; virtual reality
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (G1) (Placebo Comparator): Control group (G1): in which the suit shall be switched on, but with the current of all electrodes at 0 mA.
  Interventions: Device: The Exopulse Mollii Suit on a Fibromyalgia patient
- Suit group (G2) (Experimental): Suit group (G2): will only receive treatment with the neuromodulation suit at the intensity preset by the manufacturer and according to the assessment criteria. The duration of the treatment will be 1 hour. Exopulse Molly Suit with all 58 electrodes active with an intensity of 2 milliamperes (mA) and pulse width of 30 milliseconds (ms)
  Interventions: Device: The Exopulse Mollii Suit on a Fibromyalgia patient
- Suit + VR group (G3): (Experimental): Suit + VR group (G3): the intervention on this group was carried out in the same way as the suit group. However, the session was different as the participant wore VR glasses besides wearing the suit for an hour. The patient sees the same room he is in and a person performing a series of exercises he must follow as indicated by the video by video and voice commands. As exercise are performed in a laying position the patient must stay in this position for the whole session.
  Interventions: Device: The Exopulse Mollii Suit on a Fibromyalgia patient
- Exercise group (G4): (Experimental): Exercise group: The procedure carried out is the same as in the suit group, but the session performed was a 1-hour session of strength exercise carried out by a certified professional.
  Interventions: Device: The Exopulse Mollii Suit on a Fibromyalgia patient

INTERVENTIONS:
Device: The Exopulse Mollii Suit on a Fibromyalgia patient — The present study consists of a comparative, randomized, controlled and clinical trial conducted to explore and compare the acute and chronic effects a treatment session with the Exopulse Mollii Suit, a treatment session with the Exopulse Mollii Suit combined with VR and a training session have on a Fibromyalgia patient.
  Other Names: a treatment session with the Exopulse Mollii Suit combined with VR on a Fibromyalgia patient; a training session have on a Fibromyalgia patient

SUMMARY:
INTRODUCTION: Fibromyalgia is a chronic condition of generalised pain that entails significant limitations in daily and social life due to pain, fatigue, sleep disturbances and mood alterations. Rehabilitation programmes try to alleviate the symptoms and seek intervention methodologies that contribute to improving the quality of life and reduce the socio-economic cost. Innovation, technology and new neurophysiologically based therapeutic interventions are being integrated into rehabilitation clinics and although there are foundations and research into the potential benefits that can be obtained, research is still needed to determine intervention protocols that are more effective and efficient. The company XXX has state-of-the-art technology and equipment in order to be able to offer high quality and professional services in Extremadura and is motivated to participate in scientific, innovation and development projects in order to analyse and take advantage of the great potential of the equipment and thus offer it to society. OBJECTIVE: this project aims to compare the influence of the use of immersive virtual reality combined with Exopulse neuromodulation suits on patients with fibromyalgia. METHODOLOGY: a clinical trial is proposed with probabilistic random assignment in three groups, a control group (G1) in which patients will wear the suit on, but it will not emit any type of current. A suit group (G2), in which only the neuromodulation suit will be used, and an experimental group (G3) in which, in addition to the neuromodulation suit, virtual reality glasses will be used in full immersive mode. The variables to be analysed are: pain, postural stability, muscle activity, muscle oxygenation, thermographic distribution, heart rate variability, stress, anxiety. The acute effects will be analysed after one intervention session (pre-post intervention of one session) and the effects after a programme of 8 sessions. RESOURCES: The intervention equipment will be provided by the company and the assessment equipment by the research group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosis of fibromyalgia at least 3 months in advance.
* Minimum perceived pain intensity of 3/10 according to the Numeric Pain Rating Scale.

Exclusion Criteria:

* Having received physiotherapy 4 weeks prior to data collection.
* Personal Psychological Apprehension Scale (PPAS) score greater than 37.5.
* Contraindication to the use of electrotherapy.
* Use of opioid medication that may generate changes at the level of the Autonomic Nervous System.
* Ineligibility to participate in the study for other reasons deemed appropriate by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks
  VAS (Visual analog scale)
Postural stability | 8 weeks
  Baropodometric platform Namrol
Heart rate variability | 8 weeks
  RS800CX monitor (Polar Inc., Kempele, Finland). The Kubios HRV software (v. 3.3)
Tissue oxygenation | 8 weeks
  Oximeter. Moxy-3
Thermographic distribution | 8 weeks
  Camera E85 24" LENS. TELEDYNE FLIR. FLIR E8-XT system
Muscle activity | 8 weeks
  MDurance surface electromyography.
Level of depression and anxiety | 8 weeks
  Depression Anxiety Stress Scale
Body composition | 8 weeks
  Inbody 270
Respiratory variables (forced expiratory volume in 1 second (FEV1), 6 seconds (FEV6) and the ratio of both these values (FEV1/FEV6)) | 8 weeks
  To measure the following variables a spirometry test was conducted with a Vitalograph Asma1 spirometer
Cortical arousal | 8 weeks
  Measured trough the Critical Flicker Fusion Threshold (CFFT) in a viewing chamber (Lafayette Instrument Flicker Fusion Control Unit Model 12021)
Functional test | 8 weeks
  chair stand test
Functional test | 8 weeks
  Handgrip strength test
Functional test | 8 weeks
  10m up and go test
Functional test | 8 weeks
  One leg balance
Pressure pain threshold | 8 weeks
  The algometer used was a Wagner FPKTM algometer with a blunt rubber tip of 1cm. The lateral epicondyle (2 cm distal to the epicondyles), and the inside of the knee (at the medial fat pad proximal to the joint line)
Salivary Biomarkers | 8 weeks
  Unstimulated whole saliva was collected at rest and after exercise for each participant by direct draining into an ice-cold collection tube (pre-weighted) for 3 min After saliva collection, tubes with the samples were weighted (for saliva flux evaluation, mL/min), centrifuged at 1500× g for 10 min to remove food and cell debris, and the supernatant was stored at -20 ◦C until analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandro Rubio Zarapuz, Madrid, Spain